CLINICAL TRIAL: NCT06956755
Title: Registry of Myelodysplastic Syndromes and Therapy-related Acute Myeloid Leukemia
Status: Recruiting | Type: Observational
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Responsible Party: Sponsor
Other Study IDs: GFM-MDS Registry
Record Dates: First submitted 2025-03-05; First posted 2025-05-04 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myeloid, Acute
Keywords: MDS; t-AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Registry MDS is an ongoing, observational study that has collected longitudinal data on diagnostics, demographics, clinical parameters, and health Care Interventions (HCI) from patients with MDS and therapy-related acute myeloid leukemia

DETAILED DESCRIPTION:
The Registry MDS is an ongoing, observational study that has collected longitudinal data on diagnostics, demographics, clinical parameters, and health Care Interventions (HCI) from patients with MDS and therapy-related acute myeloid leukemia.

This registry was created in July 2003 by GFM Group. It is conducted in accordance with the French law on data processing and freedom relating to the processing of personal data in the field of health (law n°78-17 of 6 January 1978 as amended). It has received the favorable opinion of the ethics committee for research and the authorization of the National Commission on Informatics and Freedoms. (CNIL) Included in the registry are all patients over 18 years of age with MDS or secondary chemo- and/or radio-induced leukemia diagnosed after July 2003.

The registry allows, after obtaining the patient's consent, the anonymous recording of his or her demographic (sex, age), epidemiological (medical and family history, exposure to toxicants), clinical, biological, cytological and cytogenetic data. Included in the registry are all patients over 18 years of age with MDS or secondary chemo- and/or radio-induced leukemia diagnosed after July 2003.

The registry allows, after obtaining the patient's consent, the anonymous recording of his or her demographic (sex, age), epidemiological (medical and family history, exposure to toxicants), clinical, biological, cytological and cytogenetic data.

To date, 70 GFM centers participate in this registry, 5300 patients have been included. Approximately 400 to 500 new patients are currently included per year.

Data are recorded and entered through the web-based e-CRF by haematology centers in 70 centers of GFM at inclusion and Follow-up of the patients every six months.

Data analyses are conducted by the SBIM (Medical and Biostatistical Computing at service of Pr Sylvie CHEVRET, Hospital Saint Louis). Data quality control including monitoring of both clinical execution and data collection implemented from the initiation of the Registry has resulted in high quality data.

Registry MDS has included the most patients and has proven itself as a well-established operational, and constantly evolving project in an elderly population.

The registration of new patients is still ongoing, and the follow-up of the project is unlimited.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age > 18 years
* Patients with myelodysplastic syndrome and therapy-related acute myeloid leukemia
* Able and willing to provide written informed consent

Exclusion Criteria:

* Age <18 years
* Patient is unwilling or unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included in the "Registry" are all patients over 18 years of age with myelodysplastic syndrome and therapy-related acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 6990 (Estimated)
Dates: Start 2003-07-07 (Actual); Primary Completion 2030-01-05 (Estimated); Study Completion 2031-01-05 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level Unit of Measure g/dL | At enrollment
  Hemoglobin concentration in patients at the time of inclusion.
Absolute neutrophil count / Unit of Measure G/L | At enrollment
  Neutrophil count measured at baseline
Platelet count Unit of Measure / Unit of Measure: %G/L | At enrollment
  Neutrophil count measured at baseline
Percentage of bone marrow blasts at enrollment / Unit of Measure: percent | At enrollment
  Proportion of blasts in bone marrow aspirate
Presence of multilineage dysplasia at enrollment / Unit of Measure percent of patients | At enrollment
  Number and proportion of patients with multilineage dysplasia
Cytogenetic abnormalities at enrollment / Unit of Measure percent of patients | At enrollment
  Distribution of cytogenetic profiles observed in patients (e.g., normal karyotype, del(5q), complex karyotype, etc.).
IPSS-R risk classification at enrollment / Unit of Measure percent of patients by category | At enrollment
  Number and proportion of patients in each IPSS-R risk category.
Presence of somatic mutations at enrollment / Unit of Measure: percent of patients | At enrollment
  o Description: Frequency of key somatic mutations (e.g., SF3B1, TP53, ASXL1, etc.) identified in included patients
Demographic characteristics at enrollment / Unit of Measure: Descriptive (e.g., mean ± SD for age, % for sex distribution) | At enrollment
  Distribution of age, sex, and other demographic parameters among included patients

SECONDARY OUTCOMES:
Overall survival | From diagnosis until death or last follow-up, up to 120 months
  Time from diagnosis to death from any cause or last follow-up Progression-free survival Bone marrow failure (anemia, neutropenia and thrombocytopenia) Treatment duration and time response Time to IPSS progression, Rate and time to AML evolution Time-to-transfusion dependency Cytogenetic and molecular response
Progression-free survival | From diagnosis until progression, AML transformation, or death, assessed up to 120 months
  Time from diagnosis to progression to higher-risk MDS, transformation to AML, or death from any cause
Incidence of bone marrow failure events (anemia, neutropenia, thrombocytopenia) | From diagnosis until last follow-up, up to 120 months
  Number of patients presenting with hemoglobin <10 g/dL, neutrophils <1.0 G/L, or platelets <100 G/L during follow-up.
Duration of first-line treatment for MDS | From treatment initiation until discontinuation or last follow-up, assessed up to 60 months
  Time from initiation to discontinuation of the first-line therapeutic regimen
Time to first documented treatment response | From treatment start to first response, assessed up to 60 months
  Time from treatment initiation to the first response according to IWG-MDS 2006 criteria.
Time to transformation to acute myeloid leukemia (AML) | From diagnosis until AML confirmation or last follow-up, up to 120 months
  Time from MDS diagnosis to confirmed AML transformation (≥20% blasts in bone marrow).
Time to transfusion dependency | From diagnosis to transfusion dependency or last follow-up, up to 120 months
  Time from diagnosis to the need for regular transfusions, defined as ≥2 units/month for ≥2 consecutive months.
Cytogenetic and molecular response rates | Assessed during follow-up, up to 120 months
  Number and proportion of patients achieving partial or complete cytogenetic and/or molecular responses during follow-up.evaluations.
Time to progression on IPSS score | From initial classification to IPSS progression or last follow-up, up to 120 months
  Time from initial IPSS classification (very low/low) to high or very high-risk category.

CONTACTS AND LOCATIONS:
Locations (1):
- Aspasia Stamatoullas, Rouen, France